CLINICAL TRIAL: NCT05218434
Title: A Randomised, Double-blind, Placebo-controlled, Study of the Safety, Tolerability, and Pharmacokinetics of AX-158 Following Administration of Single and, Multiple Ascending Oral Doses and Food Effect Sub-study in Healthy Male Volunteers
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics and Food Effect After Single and Multiple Ascending Oral Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Artax Biopharma Inc (Industry)
Collaborators: Simbec-Orion Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AX-158-101
Record Dates: First submitted 2021-12-02; First posted 2022-02-01 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part A - 5mg AX-158 (Experimental): AX-158 oral Single (Single Ascending Dose)
  Interventions: Drug: AX-158
- Part A - 10mg AX-158 (Experimental): AX-158 oral Single (Single Ascending Dose)
  Interventions: Drug: AX-158
- Part A - 15mg AX-158 or Placebo (Experimental): AX-158 oral Single (Single Ascending Dose)
  Interventions: Drug: AX-158
- Part A - 25mg AX-158 (Experimental): AX-158 oral Single (Single Ascending Dose)
  Interventions: Drug: AX-158
- Part A -50mg AX-158 (Experimental): AX-158 oral Single (Single Ascending Dose)
  Interventions: Drug: AX-158
- Part B - 15mg AX-158 Fed state (Experimental): AX-158 oral single dose with food
  Interventions: Drug: AX-158
- Part B - 15mg AX-158 Fasted (Experimental): AX-158 oral single dose without food
  Interventions: Drug: AX-158
- Part C - 5mg AX-158 (Experimental): AX-158 oral daily dose for 10 days (Multiple Ascending Dose)
  Interventions: Drug: AX-158
- Part C - 10mg AX-158 (Experimental): AX-158 oral daily dose for 10 days (Multiple Ascending Dose)
  Interventions: Drug: AX-158
- Part C - 15mg AX-158 (Experimental): AX-158 oral daily dose for 10 days (Multiple Ascending Dose)
  Interventions: Drug: AX-158
- Part A - Placebo (Experimental): Placebo oral Single (Single Ascending Dose)
  Interventions: Drug: AX-158
- Part C - Placebo (Experimental): Placebo oral daily dose for 10 days (Multiple Ascending Dose)
  Interventions: Drug: AX-158

INTERVENTIONS:
Drug: AX-158 — Oral administrations of AX-158
  Other Names: Placebo

SUMMARY:
This is a Phase I Healthy volunteer study with the primary objective to evaluate the safety and pharmacokinetics profile of AX-158. The first part will evaluate single ascending dose administrations. A substudy will be performed as well to evaluate possible impact of food on drug exposure if administered under fasted or fed state. The second part will evaluate multiple ascending dose over 10 days of dosing in fed or fast state depending on the results of the substudy food effect on AX-158.

DETAILED DESCRIPTION:
This is a phase I, randomised, double-blind , placebo controlled study to investigate the safety, tolerability, and PK of AX-158 in healthy male participants following single (Part A) and multiple (Part C) ascending doses including food effect (Part B).The study will be conducted in three parts (Part A, Part B and Part C). Part A will enrol 8 participants per cohort randomised (3 :1) to receive AX-158 (6 participants) or placebo (2 participants). Part A will follow a single ascending dose (SAD) design with all participants receiving one dose of AX-158 (or placebo) in the fasted state. Part B (Food Effect) will be conducted in 8 participants in a cross-over manner; each participant will receive AX-158 in the fed and fasted state. Part C will enrol 8 participants per cohort randomised to (3 :1) to receive AX-158 (6 participants) or placebo (2 participants). Part C will follow a multiple ascending dose (MAD) design with participants receiving AX-158 (or placebo) once daily for 10 consecutive days, in a fed or fasted state (depending on the outcome of the Part B (Food Effect).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male participant, between 18 and 50 years of age, inclusive.
2. Male participant (and partner of childbearing potential) willing to use a highly effective method of contraception in addition to a condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the participant) from first dose until 4 months after last dose of Investigational Medicinal Product (IMP).
3. Participant with a body mass index (BMI) of 18-30kg/m2. BMI = body weight (kg) / [height (m)]2.
4. Total serum bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 x upper limit of normal (ULN). If total bilirubin is above the upper limit of normal and is then fractionated, direct bilirubin must be within normal limits.
5. Total serum Testosterone levels 2 x above the lower limit of the normal range within 28 days before the first dose administration of the IMP.
6. Participant with a negative urinary drugs of abuse (DOA) screen (including alcohol) test results, determined within 28 days before the first dose administration of the IMP (N.B.: A positive test result may be repeated at the Investigator's discretion).
7. Participant with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg)) and hepatitis C virus antibody (HCV Ab) test results at Screening.
8. No clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 28 days before first dose of IMP including a QRS interval > 120ms, PR interval > 220ms and QTcF > 450ms.
9. No clinically significant abnormalities in vital signs (e.g., blood pressure/pulse rate, respiration rate and oral temperature) determined within 28 days before first dose of IMP.
10. Participant must be available to complete the study (including all follow-up visits).
11. Participant must satisfy an Investigator about his fitness to participate in the study.
12. Participant must provide written informed consent to participate in the study.
13. Participants with a negative COVID-19 PCR test on admission.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence IMP absorption.
2. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 28 days or 5 half-lives (whichever is longer) prior to the first dose of IMP. Occasional use of paracetamol will be allowed.
3. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction.
4. Clinically significant history of previous allergy / sensitivity to AX-158 or any of the excipients contained within the IMP.
5. Participant with history of autoimmune disease, cardiac disease, kidney disease or any food intolerance.
6. Participants with clinically significant abnormal test results for serum biochemistry, haematology and/or urine analyses within 28 days before the first dose administration of the IMP
7. A clinically significant history of drug or alcohol abuse (defined as the consumption of more than 14 units [for male and female participants] of alcohol a week) within the past two years.
8. Inability to communicate well with the Investigators (i.e., language problem, poor mental development, or impaired cerebral function).
9. Participation in a New Chemical Entity (NCE) clinical study within the previous 3 months or five half-lives, whichever is longer, or a marketed drug clinical study within the 30 days or five half-lives, whichever is longer, before the first dose of IMP. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
10. Donation of 450 milliliters or more blood within the 3 months before the first dose of IMP.
11. Vegans, vegetarians, or other dietary restrictions (e.g., restrictions for medical, religious, or cultural reasons, etc), which would prevent participants from consuming a high-fat breakfast or standardised meal.
12. Users of nicotine products i.e., current smokers or ex-smokers who have smoked within the 6 months prior to screening or users of cigarette replacements (i.e., e-cigarettes, nicotine patches or gums).
13. Participants who have received a COVID-19 vaccine injection within 28 days prior to the first dose of IMP.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Annelize Koch, Principal Investigator — Simbec-Orion Merthyr Tydfil CF48 4DR, United Kingdom
Locations (1):
- Simbec-Orion, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borroto A, Reyes-Garau D, Jimenez MA, Carrasco E, Moreno B, Martinez-Pasamar S, Cortes JR, Perona A, Abia D, Blanco S, Fuentes M, Arellano I, Lobo J, Heidarieh H, Rueda J, Esteve P, Cibrian D, Martinez-Riano A, Mendoza P, Prieto C, Calleja E, Oeste CL, Orfao A, Fresno M, Sanchez-Madrid F, Alcami A, Bovolenta P, Martin P, Villoslada P, Morreale A, Messeguer A, Alarcon B. First-in-class inhibitor of the T cell receptor for the treatment of autoimmune diseases. Sci Transl Med. 2016 Dec 21;8(370):370ra184. doi: 10.1126/scitranslmed.aaf2140. PMID 28003549
- [Background] Roy E, Togbe D, Holdorf AD, Trubetskoy D, Nabti S, Kublbeck G, Klevenz A, Kopp-Schneider A, Leithauser F, Moller P, Bladt F, Hammerling G, Arnold B, Pawson T, Tafuri A. Nck adaptors are positive regulators of the size and sensitivity of the T-cell repertoire. Proc Natl Acad Sci U S A. 2010 Aug 31;107(35):15529-34. doi: 10.1073/pnas.1009743107. Epub 2010 Aug 13. PMID 20709959
- [Background] Roy E, Togbe D, Holdorf A, Trubetskoy D, Nabti S, Kublbeck G, Schmitt S, Kopp-Schneider A, Leithauser F, Moller P, Bladt F, Hammerling GJ, Arnold B, Pawson T, Tafuri A. Fine tuning of the threshold of T cell selection by the Nck adapters. J Immunol. 2010 Dec 15;185(12):7518-26. doi: 10.4049/jimmunol.1000008. Epub 2010 Nov 15. PMID 21078909
- [Background] Gil D, Schamel WW, Montoya M, Sanchez-Madrid F, Alarcon B. Recruitment of Nck by CD3 epsilon reveals a ligand-induced conformational change essential for T cell receptor signaling and synapse formation. Cell. 2002 Jun 28;109(7):901-12. doi: 10.1016/s0092-8674(02)00799-7. PMID 12110186
- [Background] Juraske C, Wipa P, Morath A, Hidalgo JV, Hartl FA, Raute K, Oberg HH, Wesch D, Fisch P, Minguet S, Pongcharoen S, Schamel WW. Anti-CD3 Fab Fragments Enhance Tumor Killing by Human gammadelta T Cells Independent of Nck Recruitment to the gammadelta T Cell Antigen Receptor. Front Immunol. 2018 Jul 9;9:1579. doi: 10.3389/fimmu.2018.01579. eCollection 2018. PMID 30038626
- [Background] Borroto A, Arellano I, Blanco R, Fuentes M, Orfao A, Dopfer EP, Prouza M, Suchanek M, Schamel WW, Alarcon B. Relevance of Nck-CD3 epsilon interaction for T cell activation in vivo. J Immunol. 2014 Mar 1;192(5):2042-53. doi: 10.4049/jimmunol.1203414. Epub 2014 Jan 27. PMID 24470497
- [Background] Borroto A, Arellano I, Dopfer EP, Prouza M, Suchanek M, Fuentes M, Orfao A, Schamel WW, Alarcon B. Nck recruitment to the TCR required for ZAP70 activation during thymic development. J Immunol. 2013 Feb 1;190(3):1103-12. doi: 10.4049/jimmunol.1202055. Epub 2012 Dec 24. PMID 23267019
- [Background] Lettau M, Pieper J, Gerneth A, Lengl-Janssen B, Voss M, Linkermann A, Schmidt H, Gelhaus C, Leippe M, Kabelitz D, Janssen O. The adapter protein Nck: role of individual SH3 and SH2 binding modules for protein interactions in T lymphocytes. Protein Sci. 2010 Apr;19(4):658-69. doi: 10.1002/pro.334. PMID 20082308
- [Background] Yiemwattana I, Ngoenkam J, Paensuwan P, Kriangkrai R, Chuenjitkuntaworn B, Pongcharoen S. Essential role of the adaptor protein Nck1 in Jurkat T cell activation and function. Clin Exp Immunol. 2012 Jan;167(1):99-107. doi: 10.1111/j.1365-2249.2011.04494.x. PMID 22132889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment for this study was undertaken in South Wales in the United Kingdom. A sufficient number of participants were screened in order to successfully recruit 64 eligible participants.
Pre-assignment Details: Volunteers were screened to the inclusion/exclusion criteria of the study protocol. The following assessments were performed: Physical exam, Demographics,ECG,Vital signs, Safety Laboratory testing/Urinalysis.
Groups:
- Part A - 5 mg AX-158: Single Oral Dose of 5 mg AX-158 administered on Day 1
- Part A - 10 mg AX-158: Single Oral Dose of 10 mg AX-158 administered on Day 1
- Part A - 15 mg AX-158: Single Oral Dose of 15 mg AX-158 administered on Day 1
- Part A - 25 mg AX-158: Single Oral Dose of 25 mg AX-158 administered on Day 1
- Part A - 50 mg AX-158: Single Oral Dose of 50 mg AX-158 administered on Day 1
- Part A - Placebo Participants: Denotes participants across all Part A cohorts who received matching placebo.
- Part B - 15 mg AX-158 Fed/Fasted: Single Oral Dose of 15 mg AX-158 administered on Day 1 of treatment period 1 in the fed state following a high-fat breakfast and administered on Day 1 in a fasted state in treatment period 2.
- Part C - 5 mg AX-158: Single Oral Dose of 5 mg AX-158 administered once daily from Day 1 to Day 10
- Part C - 10 mg AX-158: Single Oral Dose of 10 mg AX-158 administered once daily from Day 1 to Day 10
- Part C - 15 mg AX-158: Single Oral Dose of 15 mg AX-158 administered once daily from Day 1 to Day 10
- Part C - Placebo: Denotes participants across all Part C cohorts who received matching placebo.
Period: Overall Study
Arm/Group | Part A - 5 mg AX-158 | Part A - 10 mg AX-158 | Part A - 15 mg AX-158 | Part A - 25 mg AX-158 | Part A - 50 mg AX-158 | Part A - Placebo Participants | Part B - 15 mg AX-158 Fed/Fasted | Part C - 5 mg AX-158 | Part C - 10 mg AX-158 | Part C - 15 mg AX-158 | Part C - Placebo
Started | 6 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 5 | 6 | 5
Completed | 6 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A - 5mg AX-158: Single Oral Dose of 5 mg AX-158 administered on Day 1
- Part A - 10mg AX-158: Single Oral Dose of 10 mg AX-158 administered on Day 1
- Part A - 15mg AX-158: Single Oral Dose of 15 mg AX-158 administered on Day 1
- Part A - 25mg AX-158: Single Oral Dose of 25 mg AX-158 administered on Day 1
- Part A - 50mg AX-158: Single Oral Dose of 50 mg AX-158 administered on Day 1
- Part A - Placebo: Denotes participants across all Part A cohorts who received matching placebo.
- Part B - 15mg AX-158 Fed/Fasted: Single Oral Dose of 15 mg AX-158 administered on Day 1 of treatment period 1 in the fed state following a high-fat breakfast and administered on Day 1 in a fasted state in treatment period 2.
- Part C - 5mg AX-158: Single Oral Dose of 5 mg AX-158 administered once daily from Day 1 to Day 10
- Part C - 10mg AX-158: Single Oral Dose of 10 mg AX-158 administered once daily from Day 1 to Day 10
- Part C - 15mg AX-158: Single Oral Dose of 15 mg AX-158 administered once daily from Day 1 to Day 10
- Total: Total of all reporting groups
Arm/Group | Part A - 5mg AX-158 | Part A - 10mg AX-158 | Part A - 15mg AX-158 | Part A - 25mg AX-158 | Part A - 50mg AX-158 | Part A - Placebo | Part B - 15mg AX-158 Fed/Fasted | Part C - 5mg AX-158 | Part C - 10mg AX-158 | Part C - 15mg AX-158 | Part C - Placebo | Total
Number analyzed (Participants) | 6 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 5 | 6 | 5 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 5 | 6 | 5 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 5 | 6 | 5 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 5 | 6 | 4 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 5 | 4 | 4 | 6 | 9 | 8 | 6 | 4 | 6 | 5 | 62
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Metres] | 1.800 (0.0620) | 1.788 (0.0370) | 1.780 (0.0594) | 1.783 (0.0699) | 1.762 (0.0436) | 1.783 (0.0532) | 1.771 (0.0617) | 1.747 (0.0592) | 1.772 (0.0694) | 1.805 (0.0485) | 1.734 (0.0488) | 1.783 (0.0513)
Weight [Mean (Standard Deviation); unit: Kg] | 83.2 (12.019) | 82.62 (5.034) | 74.60 (8.636) | 81.53 (12.829) | 75.55 (6.486) | 81.24 (10.989) | 84.34 (11.244) | 73.25 (9.194) | 76.74 (11.959) | 79.88 (12.015) | 67.78 (2.842) | 80.01 (9.638)
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.508 (2.1783) | 25.880 (2.0092) | 23.580 (2.8956) | 25.548 (2.5745) | 24.313 (1.3690) | 25.557 (3.3519) | 26.850 (3.0544) | 24.053 (3.2247) | 24.392 (3.0302) | 24.672 (4.5817) | 22.584 (1.5257) | 25.143 (2.4850)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: The number of participants with recorded treatment emergent adverse events following single and multiple doses of AX-158.
Time Frame: Up to 10 days of treatment
Measure: Number; unit: participants
Groups:
- Part B - 15 mg AX-158 Fed State; Part B - 15 mg AX-158 Fasted: Single Oral Dose of 15 mg AX-158 administered on Day 1 of treatment period 1 in the fed state following a high-fat breakfast and administered on Day 1 in a fasted state in treatment period 2.
Arm/Group | Part A - 5 mg AX-158 | Part A - 10 mg AX-158 | Part A - 15 mg AX-158 | Part A - 25 mg AX-158 | Part A - 50 mg AX-158 | Part B - 15 mg AX-158 Fed State | Part B - 15 mg AX-158 Fasted | Part C - 5 mg AX-158 | Part C - 10 mg AX-158 | Part C - 15 mg AX-158 | Part A - Placebo | Part C - Placebo
Number analyzed (Participants) | 6 | 5 | 4 | 4 | 6 | 8 | 8 | 6 | 5 | 6 | 9 | 5
participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 4

2. Secondary Outcome: Maximal Plasma Concentration (Cmax)
Description: Values calculated for derived PK parameters following samples obtained at the following timepoints:
  Part A & B:
  Day 1: pre-dose, 30 mins, 45 mins, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, Day 2: 24 hr, 36 hr, Day 3: 48 hr & Day 4: 72 hr post-Day 1 dose
  Part C:
  Day 1: pre-dose, 30 mins, 45 mins, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr post-Day 1 dose Day 2: 24 hr, 36 hr post-Day 1 dose Day 3: 48 hr post-Day 1 dose Day 4: 72 hr post-Day 1 dose Day 5: prior to dose Day 10: pre-dose, 30 mins, 45 mins, 1 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr post-Day 10 dose Day 11: 24 hr, 36 hr post-Day 10 dose Day 12: 48 hr post-Day 10 dose Day 13: 72 hr post-Day 10 dose
Time Frame: Up to 13 days following dose administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Part B - 15 mg AX-158 Fed; Part B - 15 mg AX-158 Fasted: Single Oral Dose of 15 mg AX-158 administered on Day 1 of treatment period 1 in the fed state following a high-fat breakfast and administered on Day 1 in a fasted state in treatment period 2.
Arm/Group | Part A - 5 mg AX-158 | Part A - 10 mg AX-158 | Part A - 15 mg AX-158 | Part A - 25 mg AX-158 | Part A - 50 mg AX-158 | Part B - 15 mg AX-158 Fed | Part B - 15 mg AX-158 Fasted | Part C - 5 mg AX-158 | Part C - 10 mg AX-158 | Part C - 15 mg AX-158
Number analyzed (Participants) | 6 | 5 | 4 | 4 | 6 | 8 | 8 | 6 | 5 | 6
µg/mL | 0.0831 (16.3) | 0.174 (9.7) | 0.29 (10) | 0.487 (15.8) | 0.86 (18.9) | 0.237 (20.7) | 0.273 (26.3) | 0.108 (7.1) | 0.194 (15.4) | 0.298 (17.5)

3. Secondary Outcome: Total Plasma Drug Exposure (AUC0-t)
Description: as for outcome 2
Time Frame: Up to 13 days following dose administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part A - 5 mg AX-158 | Part A - 10 mg AX-158 | Part A - 15 mg AX-158 | Part A - 25 mg AX-158 | Part A - 50 mg AX-158 | Part B - 15 mg AX-158 Fed | Part B - 15 mg AX-158 Fasted | Part C - 5 mg AX-158 | Part C - 10 mg AX-158 | Part C - 15 mg AX-158
Number analyzed (Participants) | 6 | 5 | 4 | 4 | 6 | 8 | 8 | 6 | 5 | 6
h*µg/mL | 1.07 (35.6) | 2.06 (20.8) | 3.87 (25.2) | 6.88 (34) | 11.9 (24.6) | 3.3 (36.3) | 3.43 (34) | 1.67 (22.5) | 2.65 (38.6) | 4.97 (28.5)

4. Secondary Outcome: Terminal Half Life (t1/2)
Description: as for outcome 2
Time Frame: Up to 13 days following dose administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Part A - 5 mg AX-158 | Part A - 10 mg AX-158 | Part A - 15 mg AX-158 | Part A - 25 mg AX-158 | Part A - 50 mg AX-158 | Part B - 15 mg AX-158 Fed | Part B - 15 mg AX-158 Fasted | Part C - 5 mg AX-158 | Part C - 10 mg AX-158 | Part C - 15 mg AX-158
Number analyzed (Participants) | 6 | 5 | 4 | 4 | 6 | 8 | 8 | 6 | 5 | 6
h | 8.94 (18.4) | 8.48 (13.1) | 8.56 (22.1) | 10.6 (25.4) | 9.58 (10.5) | 8.19 (25.6) | 8.44 (18.8) | 9.7 (4.7) | 8.41 (21.4) | 9.84 (20.9)

ADVERSE EVENTS:
Time Frame: Adverse Event reporting and data collection occurred over the following time frames for each study part: Part A - informed consent to follow up - up to 6 weeks Part B - informed consent to follow up - up to 8 weeks Part C - informed consent to follow up - up to 8 weeks
Description: Adverse Event and Reporting Descriptions are reported in line with definitions defined by clinicaltrials.gov
Groups:
- Part B - 15 mg AX-158 Fed: Single Oral Dose of 15 mg AX-158 administered on Day 1 of treatment period 1 in the fed state following a high-fat breakfast.
- Part B - 15 mg AX-158 Fasted: Single Oral Dose of 15 mg AX-158 administered on Day 1 in a fasted state in treatment period 2.
Arm/Group | Part A - 5 mg AX-158 | Part A - 10 mg AX-158 | Part A - 15 mg AX-158 | Part A - 25 mg AX-158 | Part A - 50 mg AX-158 | Part A - Placebo | Part B - 15 mg AX-158 Fed | Part B - 15 mg AX-158 Fasted | Part C - 5 mg AX-158 | Part C - 10 mg AX-158 | Part C - 15 mg AX-158 | Part C - Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/4 | 0/4 | 0/6 | 0/9 | 0/8 | 0/8 | 0/6 | 0/5 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/5 | 0/4 | 0/4 | 0/6 | 0/9 | 0/8 | 0/8 | 0/6 | 0/5 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/4 | 0/4 | 1/6 | 1/9 | 1/8 | 1/8 | 1/6 | 1/5 | 0/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 5 mg AX-158 (N=6) | Part A - 10 mg AX-158 (N=5) | Part A - 15 mg AX-158 (N=4) | Part A - 25 mg AX-158 (N=4) | Part A - 50 mg AX-158 (N=6) | Part A - Placebo (N=9) | Part B - 15 mg AX-158 Fed (N=8) | Part B - 15 mg AX-158 Fasted (N=8) | Part C - 5 mg AX-158 (N=6) | Part C - 10 mg AX-158 (N=5) | Part C - 15 mg AX-158 (N=6) | Part C - Placebo (N=5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — Nose Bleed
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Headache
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Hayfever
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Anxiousness
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Abdominal Bloating
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Blocked Nose
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Cough

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT05218434/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT05218434/SAP_001.pdf